CLINICAL TRIAL: NCT01966627
Title: Genetics of Fatty Liver Disease in Childhood Obesity.
Brief Title: Genetics of Fatty Liver Disease in Children
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Sonia Caprio, Principal Investigator, Yale University
Other Study IDs: 1104008388; R01HD040787 (NIH)
Record Dates: First submitted 2013-07-15; First posted 2013-10-21 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Non Alcoholic Fatty Liver Disease
Keywords: non alcoholic fatty liver; childhood obesity; genetic variants
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Pediatric Obesity | interventions — Glucose Tolerance Test; Genotype

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Subjects with DNA samples collected
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pediatric NAFLD Cohort: Overweight and obese children and adolescents at risk for non alcoholic fatty liver disease will undergo oral glucose tolerance testing (ogtt), genotyping, abdominal and liver magnetic resonance imaging (mri), and will provide a stool sample at baseline and at 2 year follow up. A small subset will undergo liver biopsy to test for hepatic steatosis and nonalcoholic steatohepatitis.
  Interventions: Other: ogtt; Other: genotyping; Other: abdominal and liver magnetic resonance imaging; Other: stool sample; Other: liver biopsy

INTERVENTIONS:
Other: ogtt — oral glucose tolerance test
Other: genotyping — genotyping to look for risk alleles
Other: abdominal and liver magnetic resonance imaging — magnetic resonance imaging scan of abdomen and liver - abdominal and liver mri
Other: stool sample — stool sample taken to investigate metabolites
Other: liver biopsy — liver biopsy to examine for cellular change and steatosis

SUMMARY:
This is a study to investigate genetic predisposition to hepatic steatosis and the expression of gluconeogenic and lipogenic genes in livers of obese children and adolescents.

Hypothesis 1: Common variants recently associated with variation in plasma TG levels identified in Genome Wide Association Studies (GWAS) (such as GCKR, PNPLA3) can affect accumulation of fat and subsequent development of Non Alcoholic Fatty Liver Disease (NAFLD). Gene variants act in additive or synergistic manner with progressive liver fat accumulation per additional risk allele.

Hypothesis 2: With increase in hepatic fat content NASH and fibrosis will increase. Furthermore, expression of lipogenic markers (SREBP1c) will increase.

DETAILED DESCRIPTION:
To establish a cohort of obese youths to prospectively analyze potential factors (genetic and nutritional factors) that might affect the expression and progression of NAFLD. This study will determine genetic markers and their ability to convey susceptibility to NAFLD in obese children and adolescents. Furthermore, potential mechanisms that might contribute to the accumulation of hepatic Triglyceride (TG) accumulation will be, for the first time, assessed by genotyping. Additionally, we will examine the presence of intestinal microbiome in the development of fatty liver through stool collection.

ELIGIBILITY:
Inclusion Criteria:

* between 7 and 18 years of age,
* overweight or obese with a BMI greater than the 85th percentile for age and gender, and
* be otherwise healthy.

Exclusion Criteria:

* the use of any medication that alters liver function, blood pressure, glucose or lipid metabolism and
* no use of any antipsychotic medication
* Youth on chronic anti-inflammatory medications or who consume alcohol are also excluded.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The majority of the research subjects will be recruited from the Yale Pediatric Obesity Clinic and the Endocrine Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 381 (Actual)
Dates: Start 2011-07; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
gene expression | Baseline
  gene mutation allele variation identification measure via gene extraction

SECONDARY OUTCOMES:
hepatic fat content | 2 years
  Abdominal MRI to measure liver fat and subcutaneous and visceral fat ratio done at baseline and 2 year follow up
glucose tolerance | 2 years
  glucose tolerance status measured by 3 hour oral glucose tolerance test done at baseline and 2 year follow up

OTHER OUTCOMES:
DNA gene sequencing of intestinal bacteria's | 2 years
  Measure microbiota diversity via stool samples to understand variance of triglycerides accumulation in liver
Use liver biopsy specimen to assess differences in gene expression, as well as inflammation. | As indicated by Pediatric Hepatolgist
  liver biopsy tissue obtained when subject is scheduled for pre-ordered biopsy by hepatologist

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Caprio, M.D., Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burgert TS, Taksali SE, Dziura J, Goodman TR, Yeckel CW, Papademetris X, Constable RT, Weiss R, Tamborlane WV, Savoye M, Seyal AA, Caprio S. Alanine aminotransferase levels and fatty liver in childhood obesity: associations with insulin resistance, adiponectin, and visceral fat. J Clin Endocrinol Metab. 2006 Nov;91(11):4287-94. doi: 10.1210/jc.2006-1010. Epub 2006 Aug 15. PMID 16912127
- [Derived] Trico D, Caprio S, Rosaria Umano G, Pierpont B, Nouws J, Galderisi A, Kim G, Mata MM, Santoro N. Metabolic Features of Nonalcoholic Fatty Liver (NAFL) in Obese Adolescents: Findings From a Multiethnic Cohort. Hepatology. 2018 Oct;68(4):1376-1390. doi: 10.1002/hep.30035. PMID 29665034